CLINICAL TRIAL: NCT05154097
Title: Immunity Duration Study Eight Years After Vaccination of Children 12 to 23 Months With the Triple Viral Vaccine (Measles, Mumps and Rubella)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Other Study IDs: ASCLIN 001/2020
Record Dates: First submitted 2020-04-14; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-09

CONDITIONS: Measles Vaccine
Keywords: Immunity duration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several studies on the duration of immunity after the vaccine try to explain the cause of susceptibility to the measles virus even after the administration of 2 doses of the viral triple vaccine, based not only on the finding of low vaccine coverage.

In the recent measles epidemic that occurred in Brazil, beginning in 2018, we verified the predominance of the D8 genotype, with different strains. The detection of these strains is an important molecular marker to define different introductions of the same genotype, in the same geographic area, enabling better knowledge and discussion of the control strategies used.

Some news circulated in the press about a possible failure of the vaccine to protect the vaccinated population against this D8 genotype.

Regarding the mumps and rubella components, analyzes of the duration of immunity will be carried out for these 2 components, in addition to measles, since the children received in 2012 the triple viral vaccine, and there are data in the literature on the drop in antibodies to mumps, over the years. For rubella, Brazil received the rubella virus elimination certificate, and the results of duration of immunity from this study, may collaborate to know the profile of duration of immunity to rubella, in this cohort vaccinated in 2012, and who is living in a period without circulation of the wild virus.

DETAILED DESCRIPTION:
In this project, the investigators propose:

* Evaluate the proportion of seropositive people for measles, mumps and rubella, in relation to the doses of the triple viral vaccine administered, and recorded on the vaccination card, and correlate with the time elapsed since the last dose, of the children vaccinated at 12 months of age, in a study carried out in 2012, and which in 2020 will be 8 or 9 years old;
* Compare antibody titers in vaccinees, at 12 - 23 months of age, in 2012, in the study that compared the mono x multidose presentations of the triple viral vaccine, evaluating the serums collected at that time, in the post-vaccination post-vaccination samples (one dose from triple viral), and stored in the biorepository, and the recent sera, from samples that will be collected in 2020, 8 years later, against the vaccine virus and the wild virus, strain D8;
* Evaluate cellular immunity to measles, rubella and mumps components, in samples collected in 2020.

Children who participated in the study in 2012 received 1 dose of the triple viral vaccine at 12 - 23 months of age. After serology, IgG, using the immunoenzymatic assay (ELISA) method, children who had not presented seroconversion to any of the components of the triple viral vaccine received another dose of the vaccine. In 2012, the PNI recommended a 2nd dose of the triple viral vaccine at 4 years of age. Probably, this year, 2020, children who are included in the study will be able to register at least 2 doses of the triple viral vaccine, at 12 months as a participant in the 2012 study, and a 2nd dose of the triple viral vaccine, if they were vaccinated. at the age of 4 as recommended by the PNI. In addition, these children may have received more doses of triple viral vaccine, if they were vaccinated in a vaccination campaign, blocking vaccination, because of the measles outbreak in Rio de Janeiro.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes, aged between 8 and 9 years and who have provenly participated in the previous 2012 study.
* Agreement by the father and / or mother, or the legal guardian, with the child's participation in the study, and signing of the Informed Consent Form (ICF) and the Informed Consent Form (TALE) by the minor.
* Willingness of the father or mother, or legal guardian, to provide name, address, telephone and other information so that they can be contacted if necessary.
* Responsible (s) able (S) to understand the risks of the experiment that, although minimal, exist.
* Child able to understand TALE and accept to participate in the study.
* Responsible to understand and sign the IC. If the guardian is not able to sign (eg illiterate), the IC can be signed by an impartial witness who has accompanied the entire procedure.
* Participation availability by performing blood collection for immunity assessment.

Exclusion Criteria:

* Refusal to collect blood.
* Skin lesions at venipuncture sites that prevent collection - in this case, postpone collection.
* Child subject to abnormal bleeding after injections.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children, aged 8 to 9 years old, who will be contacted and invited to participate in the study, and who were part of the population that participated in the previous comparative study of immunogenicity after vaccination with the triple viral.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2022-01-04 (Estimated); Primary Completion 2022-04-18 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Duration of immunity from the triple viral vaccine | 8 years after the 1st dose of measles vaccine applied in the 2012 clinical study
  The present study is expected to evaluate the duration of immunity from the triple viral vaccine over the years of life, specifically in this study in the age group of 8 to 9 years, from the capture of the cohort of vaccinated with the first dose applied to 12- 23 months in the 2012 study.

SECONDARY OUTCOMES:
proportions of seropositive individuals with an enzyme immunoassay (ELISA), such as the Geometric Average Titles for measles | 8 years after the 1st dose of measles vaccine applied in the 2012 clinical study
  Both the proportions of seropositive individuals with an enzyme immunoassay (ELISA), as well as the Average Geometric Titles for measles, are higher than those observed after vaccination at 12 to 23 months of age, according to the results found in studies previously conducted in Brazil. In this study, the analysis of the agreement between the ELISA and PRNT methods will also be performed, for the evaluation of the serology of the measles component, and the agreement of the challenge test for the vaccine and wild measles strain.

CONTACTS AND LOCATIONS:
Overall Officials: Celia Menezes Cruz, Marques, Principal Investigator — Municipal Health Secretariat of Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No